CLINICAL TRIAL: NCT04333966
Title: Parental Research on Interventions for Social Media (Project PRISM)
Brief Title: Parental Research on Interventions for Social Media
Acronym: PRISM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Texas Health Science Center (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-035; 1R34AA026332-01A1 (NIH)
Record Dates: First submitted 2020-03-30; First posted 2020-04-03 (Actual); Results first posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-09

CONDITIONS: Underage Drinking
MeSH Terms: conditions — Underage Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interactive PBI (Experimental): Parents in the interactive PBI condition will receive an interactive web-based SNS PBI with text message prompts aimed to reduce adolescent alcohol use and risky cognitions related to alcohol displays on SNS.
  Interventions: Behavioral: Interactive Social Networking Site Parent Based Intervention
- Active Control (Active Comparator): Parents in the active control condition will receive an emailed copy of the Surgeon General's Call toAction: A Guide for Families.
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: Interactive Social Networking Site Parent Based Intervention — Parents in the interactive PBI condition will receive an interactive web-based SNS PBI with text message prompts aimed to reduce adolescent alcohol use and risky cognitions related to alcohol displays on SNS.
  Arms: Interactive PBI
Behavioral: Active Control — Parents in the active control condition will receive an emailed copy of the Surgeon General's Call to Action: A Guide for Families.
  Arms: Active Control

SUMMARY:
The prevalence of underage alcohol use continues to be a public health concern. Numerous studies have reported associations between teen drinking tendencies and parental attitudes and beliefs, parental awareness of teen drinking, parental monitoring and the quality of the parent-teen relationship and communication. The extensive work in this area has resulted in parent-based intervention (PBI) efforts to prevent or reduce adolescent alcohol use. Several independent studies have indicated that teens whose parents received a PBI reported less alcohol use and fewer alcohol-related consequences. Despite these strengths, one major limitation of PBI is that they do not currently take into account the large role that social networking sites (SNS) use plays in adolescents' lives and in relation to their alcohol use. Most (90%) adolescents are on SNS, and their Facebook, Instagram, and Twitter profiles include alcohol content. Thus, adolescents are making and exposed to SNS alcohol displays and these displays are associated with high-risk drinking cognitions and alcohol use. As such, the investigators propose to develop and refine an interactive PBI designed to reduce high-risk SNS cognitions (i.e. attitudes and norms), alcohol use, and negative consequences among adolescents. To achieve study aims, the investigators propose an iterative process of focus groups in order to develop and refine the interactive PBI to be delivered in the pilot study with 1 and 6-month follow-up among 100 parent/teen dyads. The objective of this R34 application is to establish feasibility and acceptability of the newly developed interactive PBI that focuses on the role of SNS in adolescent alcohol use as well as to determine preliminary effect sizes for future studies. Determining an efficacious way to reduce alcohol use and high-risk alcohol display cognitions affords future research the opportunity to make use of social network-based interventions, thus the proposed research has great potential to serve as a catalyst for future research.

DETAILED DESCRIPTION:
Although adolescents spend an increasing amount of time with their friends, parents remain an important source of support and continue to play a key role in the lives of their adolescents. The extensive work in this area has resulted in parent based intervention (PBI) efforts to prevent or reduce adolescent alcohol use. Research has shown that teens whose parents received a PBI reported less alcohol use and fewer alcohol related consequences up to 9-month follow-up relative to controls. However, one major limitation of PBIs is that they do not currently take into account the large role that social networking sites (SNS) play in adolescents' lives and in relation to their alcohol use. Most (90%) adolescents are on SNS, and their Facebook, Instagram, and Twitter profiles include alcohol content. Thus, adolescents are making and exposed to SNS alcohol displays, and these displays are associated with high-risk cognitions and alcohol use. Research has argued that existing parental mediation techniques grounded primarily on television/film media have fundamental inadequacies when applied to more interactive media such as websites, social media, and mobile apps as they do not account for the interactivity, immersive virtual environments, and mediated communication innate to SNS. Further, most PBIs are presented in static manual form. The investigators are unaware of any study to date that has developed and tested an interactive PBI about alcohol use and the role of SNS in adolescent alcohol use. As such, the investigators propose to develop and refine an interactive PBI designed to reduce both high-risk SNS cognitions and alcohol use among adolescents. This application responds to PA-18-067 "Pilot and Feasibility Studies in Preparation for Drug and Alcohol Abuse Prevention Trials" as it aims to establish feasibility and acceptability of the newly developed interactive PBI that focuses on the role of SNS in adolescent alcohol use as well as to determine preliminary effect sizes for future studies. The specific aims are as follows: Aim 1: Develop and refine an interactive PBI targeting the influence of SNS on high-risk SNS cognitions and alcohol use among adolescents. Interactive PBI content and text message prompts will be developed through focus groups, which will inform a new interactive PBI to be tested in a pilot study (Aim 2). A total of 16 focus groups (8 parent, 8 teen) will be conducted with 8-10 people in each group with parents only being in focus groups with other parents and teens being only with other teens. Focus groups will occur in two phases whereby an initial sample of participants (4 parent and 4 teen focus groups) will engage in parent and teen specific focus groups (split by age of teen-15-17 and 18-20) in which they will be asked to view and interact with the interactive SNS PBI and generate additional PBI content. Based on focus group data from the first round of focus groups, revisions will be made for use in the remaining 8 focus groups (4 parent, 4 teen). Aim 2: Conduct a pilot study with parents and their adolescents aged 15-20 from the Dallas/Fort Worth (DFW) area to determine feasibility, acceptability, and preliminary effect sizes (to estimate power and sample size for a future R01 application). Parent/teen dyads (N=100) will be randomized to interactive PBI (n=50) or active control (n=50) with a 1- and 6-month follow-up. Parents in the interactive PBI condition will receive the interactive web-based SNS PBI with text message prompts developed and finalized through Aim 1 focus groups. Parents in the active control condition will receive an emailed copy of the Surgeon General's Call to Action: A Guide for Families. General Hypotheses (parent and teen). The investigators hypothesize that the interactive SNS PBI will be feasible (i.e., number of eligible participants, number of parents who gave consent, number of teens who gave consent, length of time to achieve planned recruitment and enrollment goal, rate of study completion and rate of study attrition) and acceptable (i.e., proportion of parents and teens who find the intervention acceptable; ease of viewing and interacting with interactive PBI content; relevance of material; finding content helpful, beneficial, important; ratings of individual web-based modules and text messages of the PBI; the proportion of parents and teens who would recommend the study to other families, and the proportion of parents and teens who found the interactive PBI to be favorable overall) relative to active control. The investigators further hypothesize that teens and parents in the interactive PBI condition will report more positive communication about alcohol and SNS at the 1- and 6-month follow-up relative to active control. Parent Hypotheses: The investigators hypothesize that at 1- and 6-month follow-up, parents in the interactive PBI condition will report greater knowledge about alcohol as well as the role of SNS in alcohol use relative to active control. Teen Hypotheses: The investigators hypothesize that teens in the interactive PBI condition will report less drinking, fewer alcohol-related negative consequences, less favorable attitudes toward posting about alcohol on SNS, greater perceived vulnerability to the risks of posting alcohol displays on SNS, and decreased normative perceptions about how many teens post alcohol displays on SNS relative to active control at 1- and 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria (Parents):

* have a child between the ages of 15-20 who currently lives with them
* believe that their child is active on at least one SNS
* live in Texas
* valid email address
* own a cell phone with text messaging capabilities and be ok with receiving messages
* provide valid contact information for their teen
* and willing to complete a 6 month long pilot study

Inclusion Criteria (Teens):

* being between the ages of 15-20
* be active on at least one SNS
* live in Texas
* valid email address
* own a cell phone with text messaging capabilities and be ok with receiving messages
* and willing to complete a 6 month long pilot study

Exclusion Criteria:

* not meeting inclusion criteria
* unwillingness to participate
* failure to provide consent (e.g., declining participation in the study)
* providing inconsistent responses (e.g., age) identified by the survey and introductory study telephone call
* and having already participated in the study as identified by overlap or consistency in computer IP addresses, contact information, and demographics.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dana M Litt, PhD, Principal Investigator — University of North Texas Health Science Center
Locations (1):
- University of North Texas Health Science Center, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No
A select number of researchers will have access to unidentified participant data at the close of the study.

REFERENCES:
- [Background] Currie, C. N. G. S., Roberts, C., Morgan, A., Smith, R., Settertobulte, W., Samdal, O., & Barnekow, V. (2012). Health policy for children and adolescents. Copenhagen: WHO Regional Office for Europe, 252.
- [Background] Steinberg, L. (2001). We know some things: Parent-adolescent relationships in retrospect and prospect. Journal of Research on Adolescence, 11(1), 1-19. doi: 10.1111/1532-7795.00001
- [Background] Steinberg L. Clinical adolescent psychology: what it is, and what it needs to be. J Consult Clin Psychol. 2002 Feb;70(1):124-8. doi: 10.1037//0022-006x.70.1.124. PMID 11860038
- [Background] Turrisi R, Padilla KK, Wiersma KA. College student drinking: an examination of theoretical models of drinking tendencies in freshmen and upperclassmen. J Stud Alcohol. 2000 Jul;61(4):598-602. doi: 10.15288/jsa.2000.61.598. PMID 10928730
- [Background] Ichiyama MA, Fairlie AM, Wood MD, Turrisi R, Francis DP, Ray AE, Stanger LA. A randomized trial of a parent-based intervention on drinking behavior among incoming college freshmen. J Stud Alcohol Drugs Suppl. 2009 Jul;(16):67-76. doi: 10.15288/jsads.2009.s16.67. PMID 19538914
- [Background] Turrisi R, Jaccard J, Taki R, Dunnam H, Grimes J. Examination of the short-term efficacy of a parent intervention to reduce college student drinking tendencies. Psychol Addict Behav. 2001 Dec;15(4):366-72. doi: 10.1037//0893-164x.15.4.366. PMID 11767270
- [Background] Turrisi R, Abar C, Mallett KA, Jaccard J. An Examination of the Mediational Effects of Cognitive and Attitudinal Factors of a Parent Intervention to Reduce College Drinking. J Appl Soc Psychol. 2010 Oct 1;40(10):2500-2526. doi: 10.1111/j.1559-1816.2010.00668.x. PMID 21318080
- [Background] Lenhart, A. (2015). Teens, Social Media & Technology Overview 2015. Pew Research Center . Retrieved from http://www.pewinternet.org/2015/04/09/teens-social-media-technology-2015/
- [Background] Cavazos-Rehg PA, Krauss MJ, Sowles SJ, Bierut LJ. "Hey Everyone, I'm Drunk." An Evaluation of Drinking-Related Twitter Chatter. J Stud Alcohol Drugs. 2015 Jul;76(4):635-43. doi: 10.15288/jsad.2015.76.635. PMID 26098041
- [Background] Moreno MA, Parks M, Richardson LP. What are adolescents showing the world about their health risk behaviors on MySpace? MedGenMed. 2007 Oct 11;9(4):9. PMID 18311359
- [Background] Moreno MA, Parks MR, Zimmerman FJ, Brito TE, Christakis DA. Display of health risk behaviors on MySpace by adolescents: prevalence and associations. Arch Pediatr Adolesc Med. 2009 Jan;163(1):27-34. doi: 10.1001/archpediatrics.2008.528. PMID 19124700
- [Background] Litt, D. Spiro, E., M., Swanson, A., & Lewis, M. A. (2018). Does Twitter referent matter?: The relationship between self versus other Twitter chatter and alcohol use and consequences among young adults. Manuscript submitted for publication.
- [Background] Litt DM, Stock ML. Adolescent alcohol-related risk cognitions: the roles of social norms and social networking sites. Psychol Addict Behav. 2011 Dec;25(4):708-13. doi: 10.1037/a0024226. Epub 2011 Jun 6. PMID 21644803
- [Background] Moreno MA, Christakis DA, Egan KG, Brockman LN, Becker T. Associations between displayed alcohol references on Facebook and problem drinking among college students. Arch Pediatr Adolesc Med. 2012 Feb;166(2):157-63. doi: 10.1001/archpediatrics.2011.180. Epub 2011 Oct 3. PMID 21969360
- [Background] Jiow, H. J., Lim, S. S., & Lin, J. (2016). Level Up! Refreshing Parental Mediation Theory for Our Digital Media Landscape. Communication Theory, 27(3), 309-328. doi:10.1111/comt.12109
- [Background] Kuntsche S, Kuntsche E. Parent-based interventions for preventing or reducing adolescent substance use - A systematic literature review. Clin Psychol Rev. 2016 Apr;45:89-101. doi: 10.1016/j.cpr.2016.02.004. Epub 2016 Mar 23. PMID 27111301
- [Background] Turrisi R, Mallett KA, Cleveland MJ, Varvil-Weld L, Abar C, Scaglione N, Hultgren B. Evaluation of timing and dosage of a parent-based intervention to minimize college students' alcohol consumption. J Stud Alcohol Drugs. 2013 Jan;74(1):30-40. doi: 10.15288/jsad.2013.74.30. PMID 23200148
- [Background] Fournier A. K., Hall E., Ricke P., Storey B. (2013). Alcohol and the social network: online social networking sites and college students' perceived drinking norms. Psychol. Popular Media Cult. 2, 86-95. 10.1037/a0032097
- [Background] Jaccard, J. and Levitz, N. (2013). Parent-based interventions to reduce adolescent problem behaviors: New directions for self-regulation approaches In G. Oettingen and P. Gollwitzer (Eds.) Self-regulation in adolescence. New York: Cambridge University Press.
- [Background] Testa M, Hoffman JH, Livingston JA, Turrisi R. Preventing college women's sexual victimization through parent based intervention: a randomized controlled trial. Prev Sci. 2010 Sep;11(3):308-18. doi: 10.1007/s11121-010-0168-3. PMID 20169410
- [Derived] Litt DM, Geusens F, Seamster A, Lewis MA. A Parent-Based Intervention for Reducing High-risk Social Media Cognitions, Alcohol Use, and Negative Consequences Among Adolescents: Protocol for a Randomized Controlled Pilot Study. JMIR Res Protoc. 2022 May 17;11(5):e38543. doi: 10.2196/38543. PMID 35579931

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only parent and teen dyads and who had both completed baseline were considered enrolled. The numbers in each milestone represent the total number of participants (parents and teens combined).
Groups:
- Interactive PBI: Parents in the interactive PBI condition will receive an interactive web-based SNS PBI with text message prompts aimed to reduce adolescent alcohol use and risky cognitions related to alcohol displays on SNS.
  Interactive Social Networking Site Parent Based Intervention: Parents in the interactive PBI condition will receive an interactive web-based SNS PBI with text message prompts aimed to reduce adolescent alcohol use and risky cognitions related to alcohol displays on SNS.
  Both parents and teens completed baseline, 1, and 6 month follow-up.
- Active Control: Parents in the active control condition will receive an emailed copy of the Surgeon General's Call toAction: A Guide for Families.
  Active Control: Parents in the active control condition will receive an emailed copy of the Surgeon General's Call to Action: A Guide for Families.
  Both parents and teens completed baseline, 1, and 6 month follow-up.
Period: Overall Study
Arm/Group | Interactive PBI | Active Control
Started (Overall number of participants who started the study by arm (parents and teens combined)) | 100 | 102
Parents Started (Parents who started the study by arm.) | 50 | 51
Teens Who Started (Teens who started the study by arm) | 50 | 51
Teen Completed (Teens who completed 6-month follow-up.) | 41 | 42
Parent Completed (Parents who completed 6 month follow-up) | 48 | 47
Completed (Overall number of participants who completed the study (6-month follow-up) by arm (parents and teens combined)) | 90 | 89
Not Completed | 10 | 13

BASELINE CHARACTERISTICS:
Population: Fully enrolled participants include those dyads where both parent and teen completed baseline. Numbers presented are for parents and teens combined (total number of participants).
Groups:
- Interactive PBI (Parents and Teens Combined): Parents in the interactive PBI condition will receive an interactive web-based SNS PBI with text message prompts aimed to reduce adolescent alcohol use and risky cognitions related to alcohol displays on SNS.
  Interactive Social Networking Site Parent Based Intervention: Parents in the interactive PBI condition will receive an interactive web-based SNS PBI with text message prompts aimed to reduce adolescent alcohol use and risky cognitions related to alcohol displays on SNS.
  Parents and teens completed both baseline, 1 month, and 6-month follow-up.
  Baseline measure sample sizes are presented for parents and teens combined for each arm.
- Control Condition (Parents and Teens Combined): Parents in the active control condition will receive an emailed copy of the Surgeon General's Call toAction: A Guide for Families.
  Active Control: Parents in the active control condition will receive an emailed copy of the Surgeon General's Call to Action: A Guide for Families.
  Parents and teens completed both baseline, 1 month, and 6-month follow-up.
  Baseline measure sample sizes are presented for parents and teens combined for each arm.
- Total: Total of all reporting groups
Arm/Group | Interactive PBI (Parents and Teens Combined) | Control Condition (Parents and Teens Combined) | Total
Number analyzed (Participants) | 100 | 102 | 202
Age, Categorical [Count of Participants; unit: Participants] — Population: Data are being reported separately for the parents and their teens/
  Participants
    Teens: number analyzed (Participants) | 50 | 51 | 101
    Teens: <=18 years | 40 | 46 | 86
    Teens: Between 18 and 65 years | 10 | 5 | 15
    Teens: >=65 years | 0 | 0 | 0
    Parents: number analyzed (Participants) | 50 | 51 | 101
    Parents: <=18 years | 0 | 0 | 0
    Parents: Between 18 and 65 years | 50 | 51 | 101
    Parents: >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data are being reported separately for the parents and their teens
  Participants
    Teens: number analyzed (Participants) | 50 | 51 | 101
    Teens: Female | 26 | 28 | 54
    Teens: Male | 24 | 23 | 47
    Parents: number analyzed (Participants) | 50 | 51 | 101
    Parents: Female | 41 | 43 | 84
    Parents: Male | 9 | 8 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data are being reported separately for parents and their teens.
  Participants
    Teens: number analyzed (Participants) | 50 | 51 | 101
    Teens: Hispanic or Latino | 16 | 33 | 49
    Teens: Not Hispanic or Latino | 32 | 15 | 47
    Teens: Unknown or Not Reported | 2 | 3 | 5
    Parents: number analyzed (Participants) | 50 | 51 | 101
    Parents: Hispanic or Latino | 13 | 33 | 46
    Parents: Not Hispanic or Latino | 37 | 18 | 55
    Parents: Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data are being reported separately for parents and their teens.
  Participants
    Parents: number analyzed (Participants) | 50 | 51 | 101
    Parents: American Indian or Alaska Native | 0 | 1 | 1
    Parents: Asian | 6 | 2 | 8
    Parents: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Parents: Black or African American | 13 | 12 | 25
    Parents: White | 29 | 31 | 60
    Parents: More than one race | 2 | 3 | 5
    Parents: Unknown or Not Reported | 0 | 2 | 2
    Teens: number analyzed (Participants) | 50 | 51 | 101
    Teens: American Indian or Alaska Native | 0 | 1 | 1
    Teens: Asian | 9 | 4 | 13
    Teens: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Teens: Black or African American | 7 | 12 | 19
    Teens: White | 26 | 28 | 54
    Teens: More than one race | 4 | 5 | 9
    Teens: Unknown or Not Reported | 4 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 100 | 102 | 0
Drinking Days per Month [Mean (Standard Deviation); unit: days] — Number of drinking days per month as reported by adolescent participants. Population: This outcome was only assessed for the teens, and thus is half of the overall enrollment number.
  days
    number analyzed (Participants) | 50 | 51 | 101
    (all) | 0.15 (0.65) | 0.22 (0.62) | 0.18 (0.63)

OUTCOME MEASURES:

1. Primary Outcome: Acceptability (Parent)- Program Usefulness
Description: Percentage of parents in the interactive PBI condition who agreed or strongly agreed that the program was useful
Time Frame: Data will be collected at 1 month follow-up
Population: Only parents in the interactive PBI condition received this item.
Measure: Count of Participants; unit: Participants
Arm/Group | Interactive PBI
Number analyzed (Participants) | 49
Participants | 42

2. Primary Outcome: Acceptability (Parent)- Relationship
Description: Percentage of parents assigned to Interactive PBI who agreed or strongly agreed that the program helped their relationship with their teen
Time Frame: Data will be collected at 1 month follow-up
Population: Only parents assigned to interactive PBI received this item
Measure: Count of Participants; unit: Participants
Arm/Group | Interactive PBI
Number analyzed (Participants) | 49
Participants | 45

3. Primary Outcome: Acceptability (Teen)- Relationship
Description: Percentage of teens assigned to interactive PBI who agreed or strongly agreed that the program helped their relationship with their parent
Time Frame: Data will be collected at 1 month follow-up
Population: Only participants assigned to interactive PBI received this item
Measure: Count of Participants; unit: Participants
Arm/Group | Interactive PBI
Number analyzed (Participants) | 47
Participants | 41

4. Primary Outcome: Acceptability (Teen)- Percentage Who Would Recommend the Program
Description: Percentage of teens assigned to the interactive PBI who would recommend the program
Time Frame: Data will be collected at 1 month follow-up
Population: Only participants assigned to interactive PBI received this item.
Measure: Count of Participants; unit: Participants
Arm/Group | Interactive PBI
Number analyzed (Participants) | 47
Participants | 45

5. Primary Outcome: Acceptability (Parent)- Percentage Who Would Recommend the Program
Description: Percentage of parents assigned to interactive PBI who would recommend the program
Time Frame: Data will be collected at 1 month follow-up
Population: Only participants assigned to interactive PBI received this item.
Measure: Count of Participants; unit: Participants
Arm/Group | Interactive PBI
Number analyzed (Participants) | 49
Participants | 45

6. Secondary Outcome: Drinking Days in Past Month (Teen)
Description: Number of drinking days in the past month.
Time Frame: Data will be collected at 1 month follow-up
Population: Only those participants who completed the 1-month follow-up were analyzed.
Measure: Mean (Standard Deviation); unit: Number of days
Arm/Group | Interactive PBI | Active Control
Number analyzed (Participants) | 45 | 46
Number of days | 0.24 (0.88) | 0.26 (0.86)

7. Secondary Outcome: Drinking Days in Past Month (Teen)
Description: Number of drinking days in the past month.
Time Frame: Data will be collected at 6 month follow-up
Population: Only participants who completed 6 month follow-up were analyzed
Measure: Mean (Standard Deviation); unit: number of days
Arm/Group | Interactive PBI | Active Control
Number analyzed (Participants) | 39 | 37
number of days | 0.18 (0.51) | 0.76 (2.36)

8. Secondary Outcome: Communication About Alcohol and Social Media (Parent)
Description: Extent to which parent spoke to teen about alcohol and social media in past month ranging from 1 = not at all to 4 = a great deal.
Time Frame: Data will be collected at 1 month follow-up
Population: All parents who completed the 1-month followup survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interactive PBI | Active Control
Number analyzed (Participants) | 50 | 51
units on a scale | 2.03 (0.68) | 1.79 (0.64)

9. Secondary Outcome: Communication About Alcohol and Social Media (Parent)
Description: Extent to which parent spoke to teen about alcohol and social media in past month from 1= not at all to 4= a great deal.
Time Frame: Data will be collected at 6 month follow-up
Population: All parents who completed 6-month followup
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interactive PBI | Active Control
Number analyzed (Participants) | 49 | 47
units on a scale | 1.80 (0.80) | 1.66 (0.66)

10. Secondary Outcome: Communication About Alcohol and Social Media (Teen)
Description: Extent to which teen spoke to teen about alcohol and social media in past month from 1= not at all to 4 = a great deal.
Time Frame: Data will be collected at 1 month follow-up
Population: All teens who completed 1-month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interactive PBI | Active Control
Number analyzed (Participants) | 49 | 48
units on a scale | 1.65 (0.68) | 1.53 (0.61)

11. Secondary Outcome: Communication About Alcohol and Social Media (Teen)
Description: Extent to which teen spoke to teen about alcohol and social media in past month from 1= not at all to 4= a great deal.
Time Frame: Data will be collected at 6 month follow-up
Population: All teens who completed 6-month follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interactive PBI | Active Control
Number analyzed (Participants) | 44 | 44
units on a scale | 1.48 (0.53) | 1.33 (0.48)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the life of study participation, which was 6 months.
Description: The definitions of adverse and serious adverse events do not differ from the clinicaltrials.gov definition. In this table, parent and teens are combined such that numbers reflect the combined sample size for parents and teens overall. We did not split by parents and teens separately as no adverse events were reported for either group in either arm. Thus, we opted to report by arm and not split by group (parent and teen).
Arm/Group | Interactive PBI | Active Control
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/102
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/102
Other Adverse Events (participants affected / at risk) | 0/100 | 0/102

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-28): https://cdn.clinicaltrials.gov/large-docs/66/NCT04333966/Prot_SAP_000.pdf